CLINICAL TRIAL: NCT05274282
Title: Use of Animation in Therapy: Effects on Symptom Levels of Children With Attention Deficit and Hyperactivity Disorder, a Randomized Trial
Brief Title: Effects of Animation Therapy on Children With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ozgun Belen, Principal Investigator, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO 15/728-22
Record Dates: First submitted 2022-02-15; First posted 2022-03-10 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Attention; Hyperactivity; Animation; Occupational Therapy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Spasm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Animation Therapy Group (Experimental): 10 sessions of Animation Therapy (1 session/week)
  Interventions: Other: Animation Therapy
- Control Group (No Intervention): No intervention

INTERVENTIONS:
Other: Animation Therapy — Stop-motion movie shooting process designed for improving attention skill and regulating hyperactive and impulsive behaviours.
  Arms: Animation Therapy Group

SUMMARY:
The aim of the study is to determine the effects of animation therapy on the main symptoms of Attention Deficit - Hyperactivity Disorder; hyperactivity, inattention and impulsivity.

DETAILED DESCRIPTION:
Attention Deficit and Hyperactivity Disorder (ADHD) is the most frequent childhood disorder, that is characterized with three main symptoms: inattention, hyperactivity, and impulsivity. Animation Therapy is the use of a stop-motion movie production process for therapeutic purposes. This new approach may have promising effect on attention because of its flow effect. Also, there is only one study on the effectiveness of Animation Therapy in literature. This study is planned to investigate the effects of Animation Therapy on the main symptoms of the disorder.

ELIGIBILITY:
Inclusion Criteria:

* Being at the age between 6-12 years.
* Being diagnosed with ADHD by a psychiatrist.
* Taking prescribed medication for treatment of ADHD.
* Having no physical, visual or mental problems.

Exclusion Criteria:

* Absence in pre- and post-intervention evaluations
* Not completing 10-weeks of re-animation approach intervention process.
* Discontinuation of medical treatment for ADHD.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Conners Parents Rating Scale-Revised Long Form | Baseline, pre-intervention
  Conners Parents Rating Scale-Revised Long Form is a 4-points-Likert-scale, consisting of 80 items. The given items are expressions defining the daily life behaviors of children at home setting due to ADHD. Parents mark a score between 0 (means "expression never suits my child's behavior) and 3 (means expression suits my child's behavior completely). It comprises of 14 behavioral categories: Oppositional, Cognitive Problems/Inattention, Hyperactivity, Anxious/Shy, Perfectionism, Social Problems, Psychosomatic, ADHD Index, Restless/Impulsive, Emotional Lability, Global Index, DSM-IV Inattention, DSM-IV Hyperactive/Impulsive, and DSM-IV Total. A higher score indicates more severe symptoms.
Conners Parents Rating Scale-Revised Long Form | Immediately after the intervention
  Conners Parents Rating Scale-Revised Long Form is a 4-points-Likert-scale, consisting of 80 items. The given items are expressions defining the daily life behaviors of children at home setting due to ADHD. Parents mark a score between 0 (means "expression never suits my child's behavior) and 3 (means expression suits my child's behavior completely). It comprises of 14 behavioral categories: Oppositional, Cognitive Problems/Inattention, Hyperactivity, Anxious/Shy, Perfectionism, Social Problems, Psychosomatic, ADHD Index, Restless/Impulsive, Emotional Lability, Global Index, DSM-IV Inattention, DSM-IV Hyperactive/Impulsive, and DSM-IV Total. A higher score indicates more severe symptoms.
Conners Teachers Rating Scale-Revised Long | Baseline, pre-intervention
  Conners Teachers Rating Scale-Revised Long is a 4-points-Likert-scale, consisting of 59 items. The items define the school life behaviors of children due to ADHD. The child's teacher marks a score from 0 (means "expression never suits child's behavior) to 3 (means expression suits child's behavior completely). It comprises 14 behavioral categories: Oppositional, Cognitive Problems/Inattention, Hyperactivity, Anxious/Shy, Perfectionism, Social Problems, ADHD Index - Inattention, ADHD Index - Hyperactivity, Restless/Impulsive, Emotional Lability, Global Index, DSM-IV Inattention, DSM-IV Hyperactive/Impulsive, and DSM-IV Total. A higher score indicates more severe symptoms.
Conners Teachers Rating Scale-Revised Long | Immediately after the intervention
  Conners Teachers Rating Scale-Revised Long is a 4-points-Likert-scale, consisting of 59 items. The items define the school life behaviors of children due to ADHD. The child's teacher marks a score from 0 (means "expression never suits child's behavior) to 3 (means expression suits child's behavior completely). It comprises 14 behavioral categories: Oppositional, Cognitive Problems/Inattention, Hyperactivity, Anxious/Shy, Perfectionism, Social Problems, ADHD Index - Inattention, ADHD Index - Hyperactivity, Restless/Impulsive, Emotional Lability, Global Index, DSM-IV Inattention, DSM-IV Hyperactive/Impulsive, and DSM-IV Total. A higher score indicates more severe symptoms.
the Scales for Diagnosing Attention-Deficit/Hyperactivity Disorder - Home Rating Scale | Baseline, pre-intervention
  the Scales for Diagnosing Attention-Deficit/Hyperactivity Disorder - Home Rating Scale measures the levels of hyperactivity, impulsivity, and inattention from the parent's perspective. It is a 4-points-Likert-scale, consisting of 40 items. Each item describes a specific behavior correlated with ADHD and parents scores items due to the frequency of behavior described by the item, considering the behaviors of the child at home setting. A high score means high frequency and more severe symptoms.
the Scales for Diagnosing Attention-Deficit/Hyperactivity Disorder - Home Rating Scale | Immediately after the intervention
  the Scales for Diagnosing Attention-Deficit/Hyperactivity Disorder - Home Rating Scale measures the levels of hyperactivity, impulsivity, and inattention from the parent's perspective. It is a 4-points-Likert-scale, consisting of 40 items. Each item describes a specific behavior correlated with ADHD and parents scores items due to the frequency of behavior described by the item, considering the behaviors of the child at home setting. A high score means high frequency and more severe symptoms.
the Scales for Diagnosing Attention-Deficit/Hyperactivity Disorder - School Rating Scale | Baseline, pre-intervention
  A scale that measures the levels of hyperactivity, impulsivity, and inattention from the teachers' perspective. It is a 4-points-Likert-scale, consisting of 39 items. Each item describes a specific behavior correlated with ADHD and parents scores items due to the frequency of behavior described by the item, considering the behaviors of the child at home setting. A high score means high frequency and more severe symptoms.
the Scales for Diagnosing Attention-Deficit/Hyperactivity Disorder - School Rating Scale | Immediately after the intervention
  A scale that measures the levels of hyperactivity, impulsivity and inattention on the perspective of the teachers. It is a 4-points-Likert-scale, consisting of 39 items. Each item describes a specific behavior correlated with ADHD and parents scores items due to frequency of behavior described by the item, considering the behaviors of the child at home setting. High score means high frequency and more severe symptom.

CONTACTS AND LOCATIONS:
Overall Officials: Özgün Belen, MSc, Principal Investigator — Kutahya Health Sciences University; Burcu Semin Akel, Professor, Study Director — İstanbul Kültür University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No